CLINICAL TRIAL: NCT04652947
Title: MR Quality + Diagnostic Performance for CHC Diagnosis - Gadoxetic Acid, Gadoteric Acid and P03277 Comparison
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018-74
Record Dates: First submitted 2020-09-09; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MRI diagnostic — no intervention, patient only have MRI

SUMMARY:
Compare diagnostic MRI performance of gadoteric acid, gadoxetic acid and P03277 for suspected CHC nodules less than 3 cm, using LIRADS criteria

ELIGIBILITY:
Inclusion Criteria:

* Patients who had all three MRI scans as part of the diagnosis of the same suspected CHC lesion(s)
* Reference diagnosis obtained for suspected CHC nodules by a diagnostic algorithm taking into account histology, imaging and follow-up

Exclusion Criteria:

* Delay between first MRI and 3rd MRI greater than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed for hepatopathy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
compare diagnostic MRI performance of gadoteric acid, gadoxetic acid and P03277 for suspected CHC nodules | 3 months
  the evaluation criteria will be the classification of each nodule according to the LiRADS citeria

IPD SHARING:
Plan to Share IPD: No